CLINICAL TRIAL: NCT01548599
Title: Shamba Maisha: Pilot Agricultural Intervention for Food Security and HIV Health Outcomes in Kenya
Acronym: Shamba
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kenya Medical Research Institute (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Shamba Maisha; R34MH094215-01 (NIH)
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: HIV; Malnutrition
Keywords: HIV; Malnutrition; Food Security; Kenya
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-sectoral agricultural intervention (Experimental): Participants enrolled at one study location will receive the Multi-sectoral agricultural intervention as specified below under the intervention.
  Interventions: Other: Multi-sectoral agricultural intervention
- Control (No Intervention): Participants enrolled at one study location will receive the standard of care. At the end of the study, participants in this arm will be eligible for the finance training and those who pay the loan down payment will be eligible for a small loan to purchase a human powered water pump, hosing, fertilizer, and certified seeds.

INTERVENTIONS:
Other: Multi-sectoral agricultural intervention — Participants in the intervention arm will receive a micro-finance loan and training on financial management and marketing skills. With the loan, each participant will receive vouchers to purchase the following items: the Money Maker hip pump, 50 feet of hosing, fertilizer, and government certified seeds. Participants in the intervention group will also receive training on the use of the Money Maker hip pump, a portable, low-cost, human-powered water pump developed by KickStart. Participants in the intervention group will also receive training from Kickstart on the use of the pump as well as complementary training in best horticultural practices.
  Arms: Multi-sectoral agricultural intervention

SUMMARY:
This pilot study aims to determine whether an agricultural intervention will improve food security, prevent treatment failure, reduce co-morbidities, and decrease secondary HIV transmission risk among people living with HIV/AIDS. The intervention will include: a) a human-powered water pump and other required farm commodities, b) a micro-finance loan (~$75) to purchase the pump and agricultural implements, and c) education in sustainable farming practices.

DETAILED DESCRIPTION:
Food insecurity and HIV/AIDS are two leading causes of morbidity and mortality in sub-Saharan Africa and are inextricably linked. Since food insecurity contributes to increased HIV transmission risk and higher HIV-related morbidity and mortality, the World Health Organization (WHO), United Nations Programme on HIV/AIDS (UNAIDS), and the World Food Programme have recommended integrating sustainable food production strategies into HIV/AIDS programming. Yet, to date there have been few studies to systematically evaluate the impact of promising food security interventions on health, economic and behavioral outcomes among people living with HIV and AIDS. To address this gap, the investigators plan to test the hypothesis that a multi-sectoral agricultural intervention delivered in Nyanza Province, Kenya will prevent highly active antiretroviral (HAART) treatment failure, reduce co-morbidities, and decrease secondary HIV transmission risk. The intervention will include: a) a human-powered water pump and other required farm commodities, b) a micro-finance loan (~$75) to purchase the pump and agricultural implements, and c) education in sustainable farming practices. To develop our intervention, th investigators have formed an interdisciplinary collaboration with organizations in the healthcare, agriculture, and microfinance sectors. Our study aims include:

1. The investigators will operationalize and pilot test key design elements of a future cluster randomized clinical trials (RCT) aimed to improve health outcomes among HAART-treated patients in Western Kenya. In conjunction with our collaborating partners, the investigators will develop the different components of the intervention, including: a) randomization procedures for cluster RCT using detailed site assessments; b) agricultural training protocols; c) procedures for control group; d) manual of operations.
2. The investigators will conduct a pilot study of an agricultural intervention to determine the preliminary impact of the intervention on mediating outcomes (food security, and household economic indicators), and on primary health outcomes of interest for the planned RCT (HIV treatment outcomes, HIV transmission risk and women's empowerment). Up to one hundred and sixty HIV-infected farmers on HAART in Western Kenya (80 at an intervention clinic and 80 at a control clinic) will be enrolled and followed for 1 year. Impacts of our intervention on mediating and primary health outcomes will be investigated separately and jointly to provide a preliminary assessment of possible direct and indirect intervention effects.
3. The investigators will assess the acceptability and feasibility of intervention and control conditions, and systematically translate lessons learned in the pilot study into the design of a cluster RCT. To accomplish Aim 3, the investigators will conduct a mixed methods process evaluation of the different intervention components and their implementation using quantitative, qualitative, and observational methods. The investigators will prepare an R01 grant for submission based on lessons learned. The ultimate goal of this work is to contribute to sustainable solutions to tackle the intersecting challenges of food insecurity, poverty, and HIV/AIDS in sub-Saharan Africa.

The ultimate goal of this work is to contribute to sustainable solutions to tackle the intersecting challenges of food insecurity, poverty, and HIV/AIDS in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* 18-49 years old
* Currently receiving HAART
* Belong to a patient support group or demonstrate willingness to join a support group.
* Have access to farming land and available surface water
* Have evidence of food insecurity, hunger and/or malnutrition (BMI<18.5 kg) based on FACES medical records during the year preceding recruitment.
* Participants must also agree to save the down payment (~$7) required for the loan, participate in the Adok Timo training.

Exclusion Criteria:

* None

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Cohen, MD, MPH, Principal Investigator — University of California, San Francisco; Sheri Weiser, MD, Principal Investigator — University of California, San Francisco; Elizabeth Bukusi, MBChB, M.Med, Principal Investigator — Kenya Medical Research Institute
Locations (2):
- Kenya (2):
  - Migori District Hospital, Migori, Nyanza
  - Rongo District Hospital, Rongo, Nyanza

REFERENCES:
- [Derived] Nicastro TM, Pincus L, Weke E, Hatcher AM, Burger RL, Lemus-Hufstedler E, Bukusi EA, Cohen CR, Weiser SD. Perceived impacts of a pilot agricultural livelihood and microfinance intervention on agricultural practices, food security and nutrition for Kenyans living with HIV. PLoS One. 2022 Dec 14;17(12):e0278227. doi: 10.1371/journal.pone.0278227. eCollection 2022. PMID 36516159
- [Derived] Butler LM, Bhandari S, Otieno P, Weiser SD, Cohen CR, Frongillo EA. Agricultural and Finance Intervention Increased Dietary Intake and Weight of Children Living in HIV-Affected Households in Western Kenya. Curr Dev Nutr. 2020 Jan 11;4(2):nzaa003. doi: 10.1093/cdn/nzaa003. eCollection 2020 Feb. PMID 31998859
- [Derived] Hatcher AM, Lemus Hufstedler E, Doria K, Dworkin SL, Weke E, Conroy A, Bukusi EA, Cohen CR, Weiser SD. Mechanisms and perceived mental health changes after a livelihood intervention for HIV-positive Kenyans: Longitudinal, qualitative findings. Transcult Psychiatry. 2020 Feb;57(1):124-139. doi: 10.1177/1363461519858446. Epub 2019 Jun 26. PMID 31242065
- [Derived] Weiser SD, Hatcher AM, Hufstedler LL, Weke E, Dworkin SL, Bukusi EA, Burger RL, Kodish S, Grede N, Butler LM, Cohen CR. Changes in Health and Antiretroviral Adherence Among HIV-Infected Adults in Kenya: Qualitative Longitudinal Findings from a Livelihood Intervention. AIDS Behav. 2017 Feb;21(2):415-427. doi: 10.1007/s10461-016-1551-2. PMID 27637497
- [Derived] Cohen CR, Steinfeld RL, Weke E, Bukusi EA, Hatcher AM, Shiboski S, Rheingans R, Scow KM, Butler LM, Otieno P, Dworkin SL, Weiser SD. Shamba Maisha: Pilot agricultural intervention for food security and HIV health outcomes in Kenya: design, methods, baseline results and process evaluation of a cluster-randomized controlled trial. Springerplus. 2015 Mar 12;4:122. doi: 10.1186/s40064-015-0886-x. eCollection 2015. PMID 25992307
- See also: Research Article on Shamba Maisha: A pilot study assessing impacts of a micro-irrigation intervention on the health and economic wellbeing of HIV patients — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2877674/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants received the multisectoral agricultural Intervention
- Control Arm: Participants received the standard of care
Period: Overall Study
Arm/Group | Intervention | Control Arm
Started | 72 | 68
Completed | 66 | 66
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Participants received the fiance and agricultural Intervention
- Total: Total of all reporting groups
Arm/Group | Intervention | Control Arm | Total
Number analyzed (Participants) | 72 | 68 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (0.8) | 38 (0.8) | 37.5 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 35 | 33 | 68
Education >= Secondary school [Count of Participants; unit: Participants] | 14 | 12 | 26
Current married [Count of Participants; unit: Participants] | 54 | 54 | 108
Number of people in household [Mean (Standard Deviation); unit: people per household] | 6 (0.2) | 7 (0.3) | 6.5 (0.2)
Severely food insecure (vs. moderately) [Count of Participants; unit: Participants] — Per the Household Food Insecurity Access Scale Indicator Guide, v.3, a moderately food insecure household sacrifices quality more frequently, by eating a monotonous diet or undesirable foods sometimes or often and/or has started to cut back on quantity by reducing the size of meals or number of meals, rarely or sometimes. A severely food insecure household has graduated to cutting back on meal size or number of meals often, and/or experiences running out of food, going to bed hungry, and/or going a whole day and night without eating, even as infrequently as rarely.
  Participants | 57 | 58 | 115
BMI < 18.5 kg/m^2 [Count of Participants; unit: Participants] | 13 | 5 | 18
Weekly food expenditures [Mean (Standard Deviation); unit: Kenyan Shillings] | 1694 (117) | 2176 (127) | 1928 (122)
Weekly nonfood expenditures [Mean (Standard Deviation); unit: Kenyan Shillings] | 5931 (1559) | 14788 (1941) | 10233 (1750)
Frequency of food consumption [Mean (Standard Deviation); unit: Times per week] | 69.6 (3.1) | 93.9 (3.2) | 81.4 (3.1)
CD4+ [Mean (Standard Deviation); unit: (cells/microlitre)] | 497 (32.7) | 536 (37.7) | 516 (35.2)
Viral load <40 copies/ml [Count of Participants; unit: Participants] | 35 | 49 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HIV Viral Load < 40 Copies/ML at 1 Year
Description: Compare the percentage of participants who achieve HIV viral suppression (defined as <40 copies/mL) at 1 year among intervention and control arms.
Time Frame: 1 year
Population: All 140 enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-sectoral Agricultural Intervention | Control
Number analyzed (Participants) | 72 | 68
Participants | 52 | 44
Statistical Analysis 1: Comparison: Multi-sectoral Agricultural Intervention vs Control; Test type: Superiority; p = 0.002, Mixed Models Analysis; Odds Ratio, log = 2.028, 95% CI 2-sided [0.766 to 3.289]

2. Primary Outcome: Change From Baseline in CD4 Count at 1 Year
Description: Compare change in cluster of differentiation 4 (CD4) count from baseline to 1 year among intervention and control arms.
Time Frame: 1 year
Population: All 140 enrolled participants
Measure: Mean (Standard Error); unit: cells/microliter
Groups:
- Intervention: Participants enrolled at one study location will receive the Multi-sectoral agricultural intervention as specified below under the intervention.
  Multi-sectoral agricultural intervention: Participants in the intervention arm will receive a micro-finance loan and training on financial management and marketing skills. With the loan, each participant will receive vouchers to purchase the following items: the Money Maker hip pump, 50 feet of hosing, fertilizer, and government certified seeds. Participants in the intervention group will also receive training on the use of the Money Maker hip pump, a portable, low-cost, human-powered water pump developed by KickStart. Participants in the intervention group will also receive training from Kickstart on the use of the pump as well as complementary training in best horticultural practices.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 72 | 68
cells/microliter | 80.74 (30.1) | -89.25 (30.1)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline in Frequency of Food Consumption at 1 Year
Description: Food frequency will be measured as the number of different foods or food groups and the frequency consumed over a given reference period, as adapted from the World Food Programme Food Consumption Score. Minimum = 0, maximum = 392. Higher scores reflect more frequent food consumption.
Time Frame: Baseline and 1 year
Population: All 140 enrolled participants
Measure: Mean (Standard Error); unit: Total times consumed/week
Arm/Group | Multi-sectoral Agricultural Intervention | Control
Number analyzed (Participants) | 72 | 68
Total times consumed/week | 9.621 (2.660) | 0.184 (2.660)
Statistical Analysis 1: Comparison: Multi-sectoral Agricultural Intervention vs Control; Test type: Superiority; p = 0.013, Mixed Models Analysis

4. Secondary Outcome: Percentage of Participants Who Engaged in Unprotected Sex With a Sero-Negative Partner at 1 Year
Description: Assess sexual risk behaviors including unprotected sex with a partner that is HIV-negative or of unknown serostatus.
Time Frame: 1 year
Population: 118 sexually active participants who completed endline data collection.
Measure: Number; unit: Percentage of participants
Arm/Group | Multi-sectoral Agricultural Intervention | Control
Number analyzed (Participants) | 54 | 64
Percentage of participants | 1.85 | 3.125
Statistical Analysis 1: Comparison: Multi-sectoral Agricultural Intervention vs Control; Test type: Superiority; p = 0.378, Mixed Models Analysis; Odds Ratio (OR) = 0.261, 95% CI 2-sided [0.013 to 5.165], Standard Error of Mean 0.398

5. Secondary Outcome: Change From Baseline in Food Insecurity at Year 1
Description: Collect and analyze measures of food insecurity as assessed by the Household Food Insecurity Access Scale (HFIAS). Minimum=9, maximum=36. A higher score means worse outcomes (i.e. greater food insecurity).
Time Frame: Baseline and 1 year
Population: All 140 enrolled participants
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 72 | 68
Units on a scale | -7.387 (0.513) | -3.702 (0.513)
Statistical Analysis 1: Comparison: Intervention vs Control Arm; Test type: Superiority; p < 0.001, Mixed Models Analysis

6. Secondary Outcome: Change From Baseline in Weekly Household Food Expenditures at Year 1
Description: Assess weekly household food expenditures in Kenyan shillings. A modification of the World Bank Living Standards Measurement Study (LSMS) questionnaire will be used to measure expenditures for food consumption.
Time Frame: 1 year
Population: All 140 participants enrolled
Measure: Mean (Standard Error); unit: Kenyan shillings/week
Arm/Group | Multi-sectoral Agricultural Intervention | Control
Number analyzed (Participants) | 72 | 68
Kenyan shillings/week | 304.0 (184.5) | 83.7 (184.5)
Statistical Analysis 1: Comparison: Multi-sectoral Agricultural Intervention vs Control; Test type: Superiority; p = 0.398, Mixed Models Analysis

ADVERSE EVENTS:
Description: We did not assess participants for serious or other adverse events, other than all-cause mortality.
Arm/Group | Intervention | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/72 | 1/68
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We could not definitively separate intervention effects from cluster-level variables with 2 communities randomized. The 12-month follow-up could not detect the full range & sustainability of effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No